CLINICAL TRIAL: NCT06477055
Title: A Prospective, Multicenter, Phase II Study Evaluating the Recurrence Gene Profiles of Adjuvant Osimertinib Therapy in Resected EGFR-Mutated Non-Small-Cell Lung Cancer
Brief Title: The Recurrence Gene Profiles of Adjuvant Osimertinib Therapy in Resected Non-Small-Cell Lung Cancer
Acronym: RAISE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Professor, Hunan Province Tumor Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-IIT0612
Record Dates: First submitted 2024-06-19; First posted 2024-06-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: EGFR; Osimertinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): All the patients were treated with osimertinib.
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Osimertinib — Osimertinib, 80mg, po, qd.

SUMMARY:
This is a phase II, prospective, multicenter, study to evaluate the recurrence gene profiles of adjuvant osimertinib therapy in resected EGFR-mutated NSCLC.

DETAILED DESCRIPTION:
This is aprospective, multicenter, phase II study to evaluate the recurrence gene profiles of adjuvant osimertinib therapy in resected EGFR-mutated NSCLC. Approximately 60 NSCLC patients with EGFR-sensitive mutations (19del, L858R) who received adjuvant osimertinib after complete resection were enrolled. The primary endpoint was to assess the recurrence gene profiles of adjuvant Osimertinib therapy. The secondary endpoint was to explore of subgroups recurrence gene profiles of different recurrence types (local /distant) after adjuvant Osimertinib therapy and to describe the diverse treatment patterns in real clinical practice after the disease progressed.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent signed;
2. Age ≥ 18 years;
3. Histologically confirmed diagnosis of non-squamous non-small cell lung cancer;
4. Patients with stage IB-IIIA (TNM 8#) NSCLC undergo confirmed radical R0 resection;
5. Confirmed EGFR sensitive-mutations (exon 19 deletions, 21 L858R point mutations) prior to adjuvant osimertinib therapy;
6. Recurrence after/on Osimertinib treatment according to RECIST 1.1;
7. NGS gene test report (tumor or blood sample) at the time of recurrence;
8. Receiving or not receiving neoadjuvant treatment before surgery.

Exclusion Criteria:

1. Patients with stage I-III NSCLC whose surgical resection cannot be confirmed;
2. Received adjuvant therapy other than that specified in the ADAURA study;
3. No NGS test report at recurrence;
4. History of other malignant tumors within 2 years;
5. Patients assessed by the investigator as unfit for enrollment, such as neurological disorders or metabolic disorders, physical examination or laboratory examination suspected that the patient has a possible disease, or has treatment-related complications High risk etc.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Recurrence gene profiles | Time from first subject dose to study completion, or up to 36 month
  To assess the recurrence gene profiles of adjuvant Osimertinib therapy

SECONDARY OUTCOMES:
Recurrence gene profiles in patients with different recurrence types (local /distant) | Time from first subject dose to study completion, or up to 36 month
  To explore of subgroups recurrence gene profiles of different recurrence types (local /distant) after adjuvant Osimertinib therapy
Subsequent treatment patterns | Time from first subject dose to study completion, or up to 36 month
  To describe the diverse treatment patterns (Osi or other EGFR TKIs，± chemo) in real clinical practice after the disease progressed

OTHER OUTCOMES:
Recurrence gene profiles per DFS difference | Time from first subject dose to study completion, or up to 36 month
  To explore the different recurrence gene profiles associated with clinical efficacy (DFS) in tumour or blood samples

IPD SHARING:
Plan to Share IPD: Undecided